CLINICAL TRIAL: NCT02239562
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of Synthetic PreImplantation Factor (sPIF) in Autoimmune Hepatitis
Brief Title: sPIF CLINICAL STUDY PROTOCOL IN AUTOIMMUNE HEPATITIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christopher O'Brien, MD (Other)
Collaborators: BioIncept LLC (Industry)
Responsible Party: Sponsor-Investigator, Christopher O'Brien, MD, Professor of Clinical Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140114; 119219 (Registry Identifier: FDA IND Number)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Autoimmune Hepatitis
Keywords: sPIF; synthetic PreImplantation Factor; Autoimmune; Liver; Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune; Hepatitis | interventions — preimplantation factor, synthetic; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- SAD sPIF 0.1 (Experimental): single ascending dose (SAD) 3 patients with normal liver function tests (LFTs) and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) as follows: Single subcutaneous (SQ) dose 0.1 mg/kg sPIF or Placebo Day 1
  Interventions: Drug: sPIF; Drug: Placebo
- SAD sPIF 0.5 (Experimental): single ascending dose (SAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) as follows: single SQ dose 0.5 mg/kg sPIF or Placebo Day 1
  Interventions: Drug: sPIF; Drug: Placebo
- SAD sPIF 1.0 (Experimental): single ascending dose (SAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) as follows: Cohort 3: single SQ dose 1.0 mg/kg sPIF or Placebo Day 1
  Interventions: Drug: sPIF; Drug: Placebo
- MAD sPIF 0.1 (Experimental): multiple ascending dose (MAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) to multiple doses of sPIF SQ (one time) 1X day for 5 consecutive days (Days 1 to 5) Cohort 1: SQ 0.1 mg/kg sPIF or Placebo Days 1-5
  Interventions: Drug: sPIF; Drug: Placebo
- MAD sPIF 0.5 (Experimental): multiple ascending dose (MAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) to multiple doses of sPIF SQ 1X day for 5 consecutive days (Days 1 to 5) Cohort 1: SQ 0.5 mg/kg sPIF or Placebo Days 1-5
  Interventions: Drug: sPIF; Drug: Placebo
- MAD sPIF 1.0 (Experimental): multiple ascending dose (MAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) to multiple doses of sPIF SQ 1X day for 5 consecutive days (Days 1 to 5) Cohort 1: SQ 1.0 mg/kg sPIF or Placebo Days 1-5
  Interventions: Drug: sPIF; Drug: Placebo

INTERVENTIONS:
Drug: sPIF
  Other Names: synthetic PreImplantation Factor
Drug: Placebo
  Other Names: Ringer's lactated solution

SUMMARY:
The purpose of this study is to study the safety and tolerability of synthetic PreImplantation Factor (sPIF) in female patients with autoimmune hepatitis. Autoimmune hepatitis is a disease where the patient's immune system produces an inappropriate immune response against their own liver. PreImplantation Factor is a substance that is secreted by viable fetuses during pregnancy. PIF apparently initiates both maternal tolerance preventing the loss/rejection of the fetus. Synthetic PIF (sPIF) successfully translates PIF endogenous properties to pregnant and non-pregnant immune disorders. sPIF was found to be effective in preclinical models of autoimmunity and transplantation (published). Specifically sPIF protected the liver against immune attack. Toxicity studies (mice, dogs) have shown that high-dose sPIF administration for 2 weeks followed by 2 weeks observation period demonstrated a high safety profile. This study will evaluate the safety, tolerability and the blood level of this synthetic version of this natural compound in the circulation.

DETAILED DESCRIPTION:
Both sPIF as well as natural PIF appears to orchestrate a complex series of cytokine effects that overall appear to cause return of proper immune function and regulation rather than a nonspecific immune suppression. PIF acts on both the innate and adaptive arms of the immune system in a dynamic, diverse and synergetic manner "per need". In the pregnancy setting, PIF maintains basal immunity required for embryo and maternal survival, and aids in tolerance for self by blocking activated T cells proliferation that would otherwise harm the embryo. The activity of PIF appears to have a dual complementary mode of action that is dependent on whether the immune system is in the basal or the stimulated immune state. The sPIF concentrations that were used are in the same range as those that are present in maternal circulation of viable pregnancy. sPIF targets three major intracellular proteins that pivotal in autoimmune control.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged from 18 to 70 years old, of non-child bearing potential (to avoid the possibility if antibodies are formed to sPIF this could put the patient at risk for future fertility)
* Females must be either

  * Postmenopausal for greater than two years,
  * Postmenopausal for less than two years with an follicle stimulating hormone (FSH) level greater > 40 million international units per milliliter (mIU/mL )
  * Or documented as surgically sterile (bilateral tubal ligation, bilateral oophorectomy or post-hysterectomy) at least three months prior to the screening evaluation
* Autoimmune hepatitis as documented by a:

  * Pretreatment score ≥15
  * Or a post-treatment score of ≥17 on the International Criteria for the Diagnosis of Autoimmune Hepatitis (Appendix 2)
* Treatment with prednisone and/or other oral, immunosuppressive drug(s) must have been stabilized for at least 6 weeks prior to screening for this study.
* Stable ALT levels with a fixed dose of their immunosuppressant medications
* Subjects do not have to have had a documented relapse after completion of an initial course of therapy
* Permitted concomitant immunosuppressant medications will include

  * Azathioprine dose equal to/or less 100 mg per day,
  * Budesonide dose equal to/or less 9 mg per day,
  * Mycophenolate mofetil equal to/or less 3000 mg per day,
  * Prednisone equal to/or less than 10 mg per day
  * Ursodeoxycholic acid equal to/or less than 1000 mg per day
* In the judgment of the Investigator, be in reasonable general health, based on review of the results of a screening evaluation (to include physical examination, measurement of vital signs, 12-lead ECG trace and the collection of blood and urine for routine clinical laboratory testing), performed no more than 30 days prior to Day 1 of study.
* Patients must agree to abstain from alcohol use during their participation in the study protocol.
* Alanine aminotransferase (ALT) levels of no more than five times the upper limit of normal (reference) range (ULN) at the screening evaluation.
* Normal renal function as determined by a serum creatinine
* A female of childbearing potential who is documented as either surgically sterile (bilateral tubal ligation, bilateral oophorectomy or post-hysterectomy at least 3 months prior to the screening evaluation) or post-menopausal for ≥ 2 years.

Exclusion Criteria:

* Any other forms of chronic liver disease.
* Decompensated liver disease defined on the basis of any one of the following laboratory parameters at the screening evaluation: total bilirubin > 1.5 × ULN, prothrombin time > 1.2 × ULN, platelets ≤ 100,000/mm3, or albumin < 3 g/dL OR current or prior history of clinical hepatic decompensation (e.g., ascites, jaundice, encephalopathy or variceal hemorrhage).
* Hemoglobin < 11 g/dL at the screening evaluation.
* Serological evidence of infection with HIV upon review of the medical record.
* Evidence of hepatocellular carcinoma (i.e., screening α-fetoprotein > 50 ng/mL or other standard of care measure).
* Subjects with, or a history of clinically significant oncologic, pulmonary, hepatic, gastrointestinal, renal, other cardiovascular, hematologic, metabolic, endocrine, neurologic, immunologic or hematologic illness or any other major medical disorder that, in the judgment of the Investigator, would interfere with subject treatment, assessment or compliance with the protocol or should otherwise preclude their participation in this trial.
* Have received therapy with potentially hepatotoxic drugs within 3 months (90 days) prior to Day 1 or are expected to receive such therapy during the study.
* Patient who are expected to receive a change in their immunosuppressant therapies during the protocol.
* Patients who may receive chemotherapeutic agents (e.g., corticosteroids, immunoglobulins and other immune- or cytokine-based therapies) during the study for any other medical condition.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B. O'Brien, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Center for Liver Diseases; University of Miami, Miami, Florida
  - Chief Scientist, BIOINCEPT, LLC / Chairman, (SIEP) / Director, Ob&Gyn CAMcare Health Center, Cherry Hill, New Jersey

IPD SHARING:
Plan to Share IPD: No
There is no plan to share with other researchers.

REFERENCES:
- [Derived] Di Simone N, Di Nicuolo F, Marana R, Castellani R, Ria F, Veglia M, Scambia G, Surbek D, Barnea E, Mueller M. Synthetic PreImplantation Factor (PIF) prevents fetal loss by modulating LPS induced inflammatory response. PLoS One. 2017 Jul 12;12(7):e0180642. doi: 10.1371/journal.pone.0180642. eCollection 2017. PMID 28704412
- [Derived] Barnea ER, Vialard F, Moindjie H, Ornaghi S, Dieudonne MN, Paidas MJ. PreImplantation Factor (PIF*) endogenously prevents preeclampsia: Promotes trophoblast invasion and reduces oxidative stress. J Reprod Immunol. 2016 Apr;114:58-64. doi: 10.1016/j.jri.2015.06.002. Epub 2015 Jul 21. PMID 26257082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: sPIF (0.1, 0.5, or 1.0 mg/kg) given single SQ for 5 consecutive days. In SAD, n=18 randomized in a 2:1 sPIF/placebo ratio. 9 patients normal liver function and 9 abnormal liver function. In MAD, n=18 randomized in a 2:1 sPIF/placebo ratio. 9 patients normal liver function and 9 abnormal liver function. N=36 completed the study. total screened 36
Groups:
- SAD sPIF 0.1; SAD sPIF 0.5; SAD sPIF 1.0: single ascending dose (SAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) as follows: Single SQ dose 0.1 mg/kg sPIF or Placebo Day 1
- MAD sPIF 0.1; MAD sPIF 0.5; MAD sPIF 1.0: multiple ascending dose (MAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) to multiple doses of sPIF SQ 1X day for 5 consecutive days (Days 1 to 5) Cohort 1: SQ 0.1 mg/kg sPIF or Placebo Days 1-5
Period: Overall Study
Arm/Group | SAD sPIF 0.1 | SAD sPIF 0.5 | SAD sPIF 1.0 | MAD sPIF 0.1 | MAD sPIF 0.5 | MAD sPIF 1.0
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Females only
Groups:
- SAD sPIF 1.0: single ascending dose (SAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug:placebo) as follows: Single SQ dose 1.0 mg/kg sPIF or Placebo Day 1
- MAD sPIF 0.1: multiple ascending dose (MAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug : placebo) to multiple 0.1 mg/kg sPIF doses of sPIF administered subcutaneously once a day for 5 consecutive days (Days 1 to 5)
- MAD sPIF 0.5: multiple ascending dose (MAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug : placebo) to multiple 0.5 mg/kg sPIF doses of sPIF administered subcutaneously once a day for 5 consecutive days (Days 1 to 5)
- MAD sPIF 1.0: multiple ascending dose (MAD) 3 patients with normal LFTs and 3 patients with abnormal LFTs randomized in a 2:1 ratio (active drug : placebo) to multiple 1.0 mg/kg sPIF doses of sPIF administered subcutaneously once a day for 5 consecutive days (Days 1 to 5)
- Total: Total of all reporting groups
Arm/Group | SAD sPIF 0.1 | SAD sPIF 0.5 | SAD sPIF 1.0 | MAD sPIF 0.1 | MAD sPIF 0.5 | MAD sPIF 1.0 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 4 | 5 | 29
  >=65 years | 1 | 1 | 1 | 1 | 2 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 59 (8) | 59 (9) | 56.75 (13.40) | 58.75 (9.43) | 58.5 (7.33) | 59.25 (9.063)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 6 | 6 | 6 | 36
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Safety/Tolerability Measured by Clinical Laboratory Tests, Metabolics, Cytokines, Anti-PIF Antibody, Periodic Physical Examination, Including Vital Signs Measurements and 12-lead ECG
Description: Single Ascending Dose (SAD):
  Adverse events, concomitant medications: Days 1, 2, 3, 5, 8 Vital signs, Physical exams: Days 1, 2, 8 Complete blood counts (CBC), Serum chemistry, Liver function tests, Pharmacokinetics: Days 1, 2, 8 Lipids, Coagulation, Urinalysis, Pregnancy test: Days 1, 8 EKG, chest x-ray (CXR): Days 1 and 8
  Multiple Ascending Dose (MAD):
  Adverse events, concomitant medications: Days 1, 2, 3, 4, 5, 8, 15, 29 Vital signs, Physical exams: Days 1, 2, 3, 4, 5, 8, 15, 29 CBC, Serum chemistry, Liver function tests, Pharmacokinetics: Days 1, 3, 5, 8, 15, 29 Lipids, Coagulation, Urinalysis, Pregnancy test, EKG: Days 1, 5, 29 CXR: Days 1, 29
Time Frame: 29 Day
Population: All patients participating in each arm were assessed for adverse events by symptoms, physical examination and laboratory studies.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD sPIF 0.1 | SAD sPIF 0.5 | SAD sPIF 1.0 | MAD sPIF 0.1 | MAD sPIF 0.5 | MAD sPIF 1.0
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Liver Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Skeletal Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Muscular Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Nervous Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Endocrine Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Blood Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Skin Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Digestive Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Urinary Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Reproductive Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Liver Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Skeletal Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Muscular Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Nervous Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Endocrine Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Cardiovascular Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Blood Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Skin Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Digestive Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Urinary Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Respiratory Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  PE Reproductive Grade 2,3, or 4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Liver Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Skeletal Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Muscular Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Nervous Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Endocrine Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Cardiovascular Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Blood Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Skin Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Digestive Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Urinary Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Respiratory Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  Lab: Reproductive Grade 2,3,4 Adverse Events | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Anti-sPIF Antibodies and Drug Interactions
Description: Following sPIF administration, using a validated assay, serum samples were tested for anti-sPIF antibodies
Time Frame: 29 Day
Measure: Number; unit: participants
Arm/Group | SAD sPIF 0.1 | SAD sPIF 0.5 | SAD sPIF 1.0 | MAD sPIF 0.1 | MAD sPIF 0.5 | MAD sPIF 1.0
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
participants
  Number of Patients with anti-sPIF Antibody | 0 | 0 | 0 | 0 | 0 | 0
  Number of Patients with Drug to Drug Interactions | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected in the single ascending dose (SAD) until Day 8. Adverse events were collected in the multiple ascending dose (MAD) until Day 29. The total time period for the adverse event data collection was 26 months.
Groups:
- Single Ascending Dose Placebo: Single dose of placebo administered subcutaneously (Day 1)
- Single Ascending Dose 0.1: Single dose 0.1 mg/kg sPIF administered subcutaneously (Day 1)
- Single Ascending Dose 0.5: Single dose 0.5 mg/kg sPIF administered subcutaneously (Day 1)
- Single Ascending Dose 1.0: Single dose 1.0 mg/kg sPIF administered subcutaneously (Day 1)
- Multiple Ascending Placebo: Placebo administered subcutaneously once a day for 5 consecutive days (Days 1 to 5)
- Multiple Ascending Dose 0.1: 0.1 mg/kg sPIF administered subcutaneously once a day for 5 consecutive days (Days 1 to 5)
- Multiple Ascending Dose 0.5: 0.5 mg/kg sPIF administered subcutaneously once a day for 5 consecutive days (Days 1 to 5)
- Multiple Ascending Dose 1.0: 1.0 mg/kg sPIF administered subcutaneously once a day for 5 consecutive days (Days 1 to 5)
Arm/Group | Single Ascending Dose Placebo | Single Ascending Dose 0.1 | Single Ascending Dose 0.5 | Single Ascending Dose 1.0 | Multiple Ascending Placebo | Multiple Ascending Dose 0.1 | Multiple Ascending Dose 0.5 | Multiple Ascending Dose 1.0
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Ascending Dose Placebo (N=6) | Single Ascending Dose 0.1 (N=6) | Single Ascending Dose 0.5 (N=6) | Single Ascending Dose 1.0 (N=6) | Multiple Ascending Placebo (N=6) | Multiple Ascending Dose 0.1 (N=6) | Multiple Ascending Dose 0.5 (N=6) | Multiple Ascending Dose 1.0 (N=6)
liver fullness (bloating) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — liver fullness
transient skin irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — transient headache

LIMITATIONS AND CAVEATS:
Due to the small number of subjects, formal statistical analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less